CLINICAL TRIAL: NCT02402179
Title: Application of the Indicator Amino Acid Oxidation Technique for the Determination of Metabolic Availability of Tryptophan From White Maize Protein, in Young Adult Men
Brief Title: Metabolic Availability of Tryptophan From White Maize
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Assistant Professor, Faculty of Kinesiology and Physical Education, U of Toronto; Project Investigator, Research Institute The Hospital for Sick Children, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1000048461
Record Dates: First submitted 2015-03-19; First posted 2015-03-30 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: protein quality
MeSH Terms: interventions — Tryptophan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tryptophan Amino Acid (Experimental): 13.2, 26.4, 39.7, 52.9% of the mean tryptophan requirement of 3.78 mg/kg/d will be given to subjects.
  Interventions: Other: Tryptophan

INTERVENTIONS:
Other: Tryptophan — Tryptophan will be supplied at 13.2, 26.4, 39.7, or 52.9% of requirement; sourced from crystalline amino acid and white cornmeal maize.

SUMMARY:
Our objective is to determine the metabolic availability of Tryptophan in white maize using the indicator amino acid oxidation (IAAO) technique in adult men.

DETAILED DESCRIPTION:
Our objective is to determine the metabolic availability of Tryptophan in white maize. Seven young, healthy, male adults will receive graded levels (13.2, 26.4, 39.7, 52.9) of tryptophan requirement of 3.78 mg/kg/d as a crystalline amino acid (AA) mixture and a porridge of white cornmeal protein respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult males (20-49years old).
* Stable body weight
* Not on any medications that could affect protein and amino acid metabolism e.g. steroids.

Exclusion Criteria:

* Recent weight loss within the last 3 months or on weight reducing diet.
* Unwillingness to participate or unable to tolerate the diet.

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Metabolic Availability of Tryptophan in Corn | 9 hours
  The quality of corn protein will be assessed by measuring the amount of its tryptophan available for protein synthesis (metabolic availability) using the slope ration method. The oxidation of the indicator amino acid phenylalanine will be measured in response to feeding graded intakes of tryptophan in a reference protein patterned after egg protein, and provided as a crystalline amino acid mixture. The pattern of oxidation of phylalanine in response to tryptophan provided in corn will be compared to the pattern of oxidation obtained from feeding the reference protein. On each study day, subjects will be fed 8 hourly meals and breath samples will be taken to measure the oxidation of phenylalanine. Samples will be collected at baseline after the fourth meal, and half hourly, beginning 2.5 hrs after the 5th meal. Breath samples will be analyzed for 13CO2 enrichment.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pencharz, MD, PhD,, Principal Investigator — Senior Scientist
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Rafii M, Elango R, Ball RO, Pencharz PB, Courtney-Martin G. Metabolic Availability of the Limiting Amino Acids Lysine and Tryptophan in Cooked White African Cornmeal Assessed in Healthy Young Men Using the Indicator Amino Acid Oxidation Technique. J Nutr. 2018 Jun 1;148(6):917-924. doi: 10.1093/jn/nxy039. PMID 29741697